CLINICAL TRIAL: NCT05012748
Title: The Effects of Ketogenic Diet on the Cardiac Substrate Metabolism and Brain Perfusion
Brief Title: The Effects of Ketogenic Diet on the Heart and Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1-10-72-232-18
Record Dates: First submitted 2021-06-21; First posted 2021-08-19 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2021-06

CONDITIONS: Ketogenic Dieting
Keywords: Ketogenic dieting; Heart metabolism; Brain perfusion
MeSH Terms: interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: The study will be performed as a randomized, placebo-controlled crossover study in 12 healthy obese patients (BMI: 28-40 kg/m2) in the age group 50-70 years. Each participant will undergo two periods of three weeks, during which they must follow a ketogenic diet or a standard diet in random order with one week of wash out between periods. At the end of each period, a study day with Metabolic and PET examinations will be performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic diet (Experimental): The participants are instructed to follow a ketogenic diet consisting of 75% fat, 20% protein and 5% carbohydrates. The diet will be standardised and matched to the energy consumption of each participant.
  Interventions: Other: Ketogenic diet
- Normal western diet (No Intervention): The participants are instructed to follow a normal western diet without emphasising any particular macronutrient.

INTERVENTIONS:
Other: Ketogenic diet — The ketogenic diet will consist of 75% fat, 20% protein and 5% carbohydrates. The diet will be standardised and matched to the energy consumption of each participant. The diet does not dictate time of consumptions. The food regime will be strictly followed every day for 3 weeks, where the investigator will contact the participants every day to secure adherence.
  Arms: Ketogenic diet

SUMMARY:
A ketogenic diet consists of a high intake of fats and a limited intake of carbohydrates, which causes an increased level of ketone bodies in the body. In recent years, it has been shown that the diet has cardiovascular protective effects. The investigators have also shown that ketone bodies act as super-gasoline for the heart. In addition, an increased level of ketone bodies will improve memory and comprehension in humans, possibly due to increased blood flow in the brain.

The purpose of the experiment is to investigate how a ketogenic diet affects the heart and brain. The theory is that an increased level of ketone bodies will improve energy utilization in the heart by reducing oxygen deficiency in the heart as well as increasing blood flow in the brain.

The study participants must go through two periods of 3 weeks, during which they must eat an ordinary Danish diet and a ketogenic diet, respectively. The periods end with an examination day, where blood samples and samples from muscle and fat tissue are taken. They will also be scanned with CT, PET and MRI scans to determine their body's ability to absorb sugar, fat and ketone bodies. The investigators expect the results to be of crucial importance for dietary recommendations for people at risk for cardiovascular disease and type 2 diabetes.

DETAILED DESCRIPTION:
Background:

The ketogenic diet has long been used in the treatment of treatment-resistant epilepsy due to an unexplained but markedly reducing effect on the number of epileptic cases. In recent years, there has also been an increased focus on the potential of ketone bodies in the treatment of cardiovascular disease, however, the effect of a persistently elevated level of circulating ketone bodies (ketosis) has not been sufficiently elucidated. Ketone bodies are produced in the liver at high levels of fatty acids, and act as an important source of energy for the brain and heart during fasting. Energy production by ketone metabolism is less oxygen-intensive than both glucose and fatty acid metabolism, and ketone substances can therefore be a highly energy-efficient substrate for the heart. Insulin-resistant individuals and people with heart disease have difficulty burning glucose in the heart due to the insulin-resistant condition and are therefore dependent on other energy sources such as free fatty acids and ketones. Because ketones are oxygen-sparing compared to fatty acids, a ketogenic diet can potentially reduce the heart's need for oxygen in patients with narrowed coronary arteries.

A recent study has shown that ketone bodies are efficiently absorbed by the heart despite maximal stimulation with insulin and glucose. In the study, healthy subjects increased the level of circulating ketone bodies to approximately 4 millimolar (mM) with a continuous ketone infusion, which resulted in a 50% reduction in cardiac glucose consumption. Since the consumption of free fatty acids in the experiment was unchanged and the overall work of the heart was the same, up to 50% of the heart's energy consumption was thus covered by ketone bodies. In addition, the high levels of ketone bodies led to a marked increase in the blood flow to the heart.

Classic ketogenic diets contain 3-4 times as many grams of fat as the total amount of carbohydrate and protein. The ketone substance level is increased to approximately 7 mM compared to ~ 0.1 mM in people who eat a "regular diet". Unfortunately, the diet requires a complete dedication to the diet plan and can lead to unpleasant gastrointestinal side effects, so there are major challenges in maintaining the diet over time.

A modified ketogenic diet is therefore of great interest, where fat contributes approximately 65% of the total amount of energy consumed and the circulating ketone bodies are increased to approximately 0.4 mM after three weeks of dietary intervention. It is not yet known how high ketone levels are required to achieve a clinically protective effect in the body's vital organs, but ketone levels are expected to reach the same level as patients treated with the antidiabetic drugs, sodium-glucose cotransporter (SGLT)-2 inhibitors. SGLT-2 inhibition has in recent studies shown impressive cardiovascular and renal protective effects in type 2 diabetics, which is attributed by a number of researchers and clinicians to the effect on the elevated level of circulating ketone bodies. An increased level of ketone bodies has also been shown to improve cognitive function in patients with impaired cognition or mild Alzheimer's disease. This can potentially be explained by an increased perfusion in the blood vessels of the brain, which is seen in ketosis.

Positron Emissions Tomography (PET) combined with a computed tomography (CT) scan is a non-invasive imaging modality that is well established in oncological staging and treatment monitoring. The technique is also suitable for tracking the fate of metabolites, as most substances or metabolites can be labeled by a suitable PET isotope. PET has sufficient spatial and temporal resolution to enable direct quantification of e.g. absorption and oxidation rates, and it has been successfully used by our department to assess cardiac efficiency, oxygen consumption , and fatty acid metabolism . The investigators are currently developing and validating a PET tracer for ketone bodies called 11C-Hydroxybutyrate (11C-3-OHB) for human studies. Once developed, the investigators will be able to detect changes in the biodistribution and kinetics of ketone bodies during both a ketogenic and a standard Western diet.

Purpose:

The overall aim of the project is to investigate whether a relatively simple and inexpensive modified ketogenic diet can be an effective non-pharmacological treatment of type 2 diabetes and other people at risk for ischemic heart disease. Using non-invasive imaging at PET, the investigators want to investigate whether the metabolism of ketones and fatty acids changes as well as whether blood flow increases in the heart during ketosis. Blood and tissue samples from skeletal muscle and adipose tissue will be examined to assess the effect of the ketogenic diet on insulin sensitivity in these tissues as well as the lipid composition in the blood. In addition, the investigators will investigate whether the improved cognitive function observed with ketosis is due to an increased perfusion in the brain, which can be detected by combining 15O-water PET with a magnetic resonance (MR) scan.

Existing treatment for type 2 diabetes and ischemic heart disease often involves significant pharmacological intervention, with participants often having difficulty adhering to the correct treatment. This may be due to non-compliance, but also due to the possible interactions and side effects that pharmacological treatment may cause, especially in case of serious illness.

With the project, the investigators want to utilize state-of-the-science PET/CT heart examinations in a clinical context. The investigators therefore hope that the project highlights the possibility that a relatively simple ketogenic diet may be an effective non-pharmacological treatment of type 2 diabetes or other individuals at risk for heart disease.

Methods:

The study will be performed as a randomized, placebo-controlled crossover study in 12 healthy obese participants (BMI: 28-40 kg / m2) in the age group 50-70 years. Before inclusion, participants will be called in for a study, which includes a conversation about health, blood tests, measurement of height, weight, blood pressure and ECG. Each trial participant will undergo two trial periods of three weeks, during which they must follow resp. a ketogenic diet / standard diet in random order with one week of leaching between trial periods.

The participants will approximately once a week be contacted by telephone in both study periods with regard to to ensure compliance with the diet. In addition, the concentration of ketone bodies will be measured by the participants twice daily (7 am and 7 pm) with ketone strips on a hand-held glucose meter at their own home. If participants increase by <0.3 mM in ketone bodies after one week of ketogenic diet, they will drop out of the study without further follow-up.

At the end of each trial period, trial participants will be called to a trial day of PET scans and metabolic studies. For 72 hours up to the test days, subjects will be asked to avoid alcohol and strenuous physical activity. They will have their physical activity monitored with an activity meter as well as blood pressure / vascular stiffness with a 24-hour blood pressure monitor (24 hours). In addition, they will be asked to fast from kl. 21 in the evening before all trial days. After each trial period, participants will have a dual energy x-ray absorptiometry (DXA) scan and an MR scan.

ELIGIBILITY:
Inclusion Criteria:

* Age: 50-70-years old
* BMI: 28-40

Exclusion Criteria:

* All drugs that could affect the outcome
* HbA1c > 48 mmol/mol
* Known heart failure og episodes of acute myocardial infarction
* Liver disease ALAT > higher than 3 times of the normal level
* Kidney disease eGFR < 60 ml/min
* Blood donation in the last 3 months before inclusion
* Participation in other studies with radiation in the last 6 months
* Alcohol addiction

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Cardiac substrate metabolism and in perfusion in the brain | Measurements will be made after 3 weeks on each diet with a washout period in between
  The change in substrate metabolism and perfusion after a ketogenic diet compared to a standard western diet, will be measured with photon emission tomography (PET) combined with computed tomography (CT) and magnetic resonance (MR) scans. The values/units will be measured as radiation defined as radiation over time (becquerel/time). With specific PET-tracers we are able to measure absolute free fatty acid (palmitate tracer), perfusion (water tracer), energy (acetate tracer) and ketone bodies (beta-hydroxybutyrate tracer).

SECONDARY OUTCOMES:
Differences in circulating concentrations of free fatty acids, total cholesterol, glucose, andhemoglobine measured in mmol/l | Measurements will be made on a screening day and after 3 weeks on each diet with a washout period in between
  Measured in blood samples
Differences in circulating concentrations of lactate dehydrogenase, glucagon, hydroxybutyrate, gastric inhibitory peptide, and glucagon-like peptide-1, alanintransaminase, alkaline phosphatase, and erythropoietin measured in units/l | Measurements will be made on a screening day and after 3 weeks on each diet with a washout period in between
  Measured in blood samples
Differences in circulating concentrations c-reactive protein measured in mg/l | Measurements will be made on a screening day and after 3 weeks on each diet with a washout period in between
  Measured in blood samples
Changes in signaling in muscle and adipose tissue | Measurements will be made after 3 weeks on each diet with a washout period in between
  Western blot examinations of muscle and adipose tissue biopsies
Differences in body composition and fat distribution | Measurements will be made on a screening day and after 3 weeks on each diet with a washout period in between
  Dual energy x-ray absorptiometry scans are performed to measure changes in
  Bone mineral content, fat, and lean mass measured in g
Differences in body composition | Measurements will be made on a screening day and after 3 weeks on each diet with a washout period in between
  Dual energy x-ray absorptiometry scans are performed to measure changes in
  Bone mineral density measured in g/cm^2
Insulin sensitivity | Measurements will be made after 3 weeks on each diet with a washout period in between
  The participants will be put on a hyperinsulinemic euglycemic clamp during the study day. The amount of infused glucose during the clamp will act as a measure of the participants insulin sensitivity/resistance

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus N, Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Svart M, Rittig N, Luong TV, Gopalasingam N, Vestergaard ET, Gormsen L, Sondergaard E, Thomsen HH, Gravholt CH. Three Weeks on a Ketogenic Diet Reduces Free Testosterone and Free Estradiol in Middle-Aged Obese Men and Women. J Nutr Metab. 2024 Aug 6;2024:9301369. doi: 10.1155/2024/9301369. eCollection 2024. PMID 39139216